CLINICAL TRIAL: NCT07211919
Title: Functional MRI Guided Accelerated Intermittent Theta Burst Stimulation for Chronic Post-Concussive Syndrome: A Feasibility and Efficacy Retrospective Chart Review
Brief Title: Accelerated Transcranial Magnetic Stimulation Intervention for Post-Concussion Syndrome
Status: Completed | Type: Observational
Sponsor: Cognitive FX (Industry)
Responsible Party: Sponsor
Other Study IDs: CFX2025_PCS_TMS; 25-12-393-2253 (Other: BRANY IRB)
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Post Concussive Syndrome, Chronic; Post Concussion Symptoms; Post Concussive Syndrome; Post Concussion Syndrome; Anxiety Disorder Not Otherwise Specified
Keywords: Post Concussion Syndrome; fMRI Transcranial Magnetic Stimulation; Accelerated Intermittent Theta Burst; Functional Neuroimaging
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Concussion Symptom Participants: Participants experiencing chronic or acute symptoms resulting from a mild traumatic brain injury

SUMMARY:
This study looks at the effects of accelerated intermittent theta burst stimulation (aiTBS) on patients with chronic and acute post-concussion syndrome. Each participant was treated in an outpatient setting for about 3 hours per day, over 3 days. The participants' symptom survey scores and brain scan data were then compared before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic or acute concussion symptoms

Exclusion Criteria:

* MDD, GAD, bipolar depression, PTSD, schizophrenia, metal implants in skull, pacemaker, history of seizures, epilepsy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants were primarily recruited from referrals to Neural Effects (an insurance-based acute concussion care center tied to Cognitive FX). Additional patients were recruited from word-of-mouth referrals to our clinic for concussion care.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Post-Concussion Symptom Scale (PCSS) Score | Scores taken prior to intervention, immediately post-intervention, and 1-4 weeks post-intervention
  PCSS (post-concussion symptom scale) is a 21-question Likert scale questionnaire regarding physical, cognitive, sleep, and emotional symptoms of post-concussion syndrome. Minimum score on the scale is zero, maximum score is 126. Higher score indicates more severe symptoms.
Beck Anxiety Inventory (BAI) Score | Immediately prior to treatment, after treatment, and 1-4 weeks post-treatment
  Beck Anxiety Inventory is a 21-question Likert scale questionnaire used for measuring severity of anxiety symptoms. Minimum score is zero, maximum score is 63. Higher score indicates more severe symptoms.
Beck Depression Inventory (BDI) Score | Pre-treatment, immediately post-treatment, and 1-4 weeks post-treatment.
  Beck Depression Inventory is a 21-question multiple choice self-report inventory used for measuring severity of depression. Minimum score is zero, maximum score is 63. Higher scores indicate more severe symptoms.
Functional Neurocognitive Imaging (fNCI) Score | 1-4 weeks pre-treatment, 1-4 weeks post-treatment
  The fNCI assessment protocol combines the validity of conventional neuropsychological testing standards with the reliability and objectivity of informational data output provided by fMRI. It is a scan comparing BOLD signal and blood flow from participant's brain scan against a normative database of healthy, non-injured brains. Higher scores represent further deviation from healthy baseline, with a minimum score of zero and no theoretical maximum score. Scores below 1 are within healthy range.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Allen, PhD, Principal Investigator — Cognitive FX
Locations (1):
- Cognitive FX TMS Clinic, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared unless other researchers sign a data use agreement outlining a plan to use IPD that does not include any form of identifiable PHI.